CLINICAL TRIAL: NCT01773473
Title: Comparison Between Low Mixed Insulin and Mid Mixed Insulin AS Starter Insulin For Patients With TYpe 2 Diabetes Mellitus (CLASSIFY Study)
Brief Title: Comparison of Insulin Mix25 Versus Mix50
Acronym: CLASSIFY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14675; F3Z-CR-IOQI (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin lispro, isophane insulin lispro drug combination (25:75)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro Mix25 (Experimental): Insulin Lispro Mix25 administered subcutaneously (SC) using prefilled pen twice daily for 26 weeks.
  Interventions: Drug: Insulin Lispro Mix25
- Insulin Lispro Mix50 (Experimental): Insulin Lispro Mix50 administered SC using prefilled pen twice daily for 26 weeks.
  Interventions: Drug: Insulin Lispro Mix50

INTERVENTIONS:
Drug: Insulin Lispro Mix25 — Administered SC
  Other Names: LY275585-75
  Arms: Insulin Lispro Mix25
Drug: Insulin Lispro Mix50 — Administered SC
  Other Names: LY275585-50
  Arms: Insulin Lispro Mix50

SUMMARY:
The purpose of this study is to determine the efficacy and safety of insulin Lispro Mix25 (LM25) compared to insulin Lispro Mix50 (LM50) as an insulin starter in participants with Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 2 Diabetes Mellitus (T2DM) for at least 6 months
* Have been taking sulfonylureas, biguanide, thiazolidinedione, alpha-glucosidase inhibitor, glinide, or dipeptidyl peptidase IV inhibitor, or any combination of these
* Have a qualifying hemoglobin A1c (HbA1C) value ≥7.0% and ≤11.0% at screening
* Have a body mass index (BMI) ≥18.5 and <35.0 kilogram per square meter (kg/m²)
* Have given written informed consent to participate in the study in accordance with local regulations and the ethical review board (ERB) governing the study site

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes
* Have had more than 1 episode of severe hypoglycemia within the 6 months before screening
* Have any of the following cardiovascular conditions within 3 months prior to screening: acute myocardial infarction, New York Heart Association (NYHA) class III or class IV heart failure, or cerebrovascular accident (stroke)
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine aminotransferase levels ≥3.0 times the upper limit of the reference range at screening, as determined by the central laboratory
* Have an estimated creatinine clearance (CrCl), Cockcroft-Gault formula <30 milliliter per minute (mL/min), as determined by the central laboratory at screening
* Have evidence of a significant, active, uncontrolled endocrine or autoimmune abnormality, as judged by the investigator
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy for <5 years
* Have any other condition (such as, known drug or alcohol abuse or a psychiatric disorder) that may prevent the participants from following and completing the protocol
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- China (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ürümqi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhengzhou
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeju Special Self-Governing Pr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep

REFERENCES:
- [Derived] Su Q, Liu J, Li P, Qian L, Yang W. Relative Contribution of Fasting and Postprandial Blood Glucose in Overall Glycemic Control: Post Hoc Analysis of a Phase IV Randomized Trial. Diabetes Ther. 2018 Jun;9(3):987-999. doi: 10.1007/s13300-018-0403-7. Epub 2018 Mar 24. PMID 29574635

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 26-week treatment period (12-week, weekly-intensive, dose-adjustment period and 14-week maintenance period).
Period: Overall Study
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Started | 207 | 196
Received at Least 1 Dose of Study Drug | 207 | 196
Completed | 191 | 177
Not Completed | 16 | 19
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 0 | 4
Not completed — Physician Decision | 3 | 5
Not completed — Sponsor Decision | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-Compliance with study drug | 1 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Insulin Lispro Mix25: Insulin Lispro Mix25 administered SC using prefilled pen twice daily for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50 | Total
Number analyzed (Participants) | 207 | 196 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.74 (10.026) | 57.34 (9.664) | 56.52 (9.871)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 77 | 153
  Male | 131 | 119 | 250
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 192 | 182 | 374
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 14 | 29
  Japan | 88 | 84 | 172
  China | 80 | 76 | 156
  Korea, Republic of | 24 | 22 | 46
Duration of Type-2 Diabetes Mellitus (T2DM) [Mean (Standard Deviation); unit: years] | 9.74 (6.169) | 9.15 (6.336) | 9.45 (6.250)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26
Description: HbA1c is the glycosylated fraction of hemoglobin A which provides an estimate of a participant's blood sugar control over a 6- to 12-week period. Least Squares (LS) means were calculated by Mixed Models Repeated Measurements (MMRM) analysis using change from baseline in HbA1c at all post baseline measurement as dependent variables, treatment, blood glucose (BG) excursion, country, visit and treatment-by-visit interaction as fixed effects, baseline HbA1c value as a covariate and participants as a random effect.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least 1 dose of study drug and analyzed according to the assigned treatment regardless of study drug dose the participant received and had baseline and Week 26 HbA1c measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 192 | 179
percentage of glycosylated hemoglobin | -1.52 [-1.66 to -1.39] | -1.69 [-1.83 to -1.55]
Statistical Analysis 1: Comparison: Insulin Lispro Mix25 vs Insulin Lispro Mix50; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.01 to 0.35]

2. Secondary Outcome: Percentage of Participants Achieving HbA1c of <7.0% or ≤6.5% Baseline Through Week 26
Description: HbA1c is the glycosylated fraction of hemoglobin A which provides an estimate of a participant's blood sugar control over a 6- to 12-week period. The percentage of participants with HbA1c <7.0% or HbA1c ≤6.5% is calculated as the number of participants with an HbA1c level of the cut-off value (<7.0% or ≤6.5%) divided by the number of participants treated, then multiplied by 100.
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least 1 dose of study drug and analyzed according to the assigned treatment regardless of study drug dose the participant received and had baseline and at least 1 post-baseline HbA1c measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
percentage of participants
  <7.0% | 45.9 | 59.7
  ≤6.5% | 26.1 | 42.3

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at Week 26
Description: LS means were calculated by MMRM analysis using change from baseline in FBG variables at all post baseline measurement as dependent variables, treatment, country, BG excursion, visit and treatment-by-visit interaction as fixed effects, baseline self-monitoring blood glucose (SMBG) variable value as a covariate and participants as a random effect.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least 1 dose of study drug and analyzed according to the assigned treatment regardless of study drug dose the participant received and had baseline and Week 26 FBG measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
millimoles per liter (mmol/L) | -2.37 [-2.68 to -2.06] | -1.99 [-2.30 to -1.68]

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: LS means were calculated by MMRM analysis using change from baseline in weight variables at all post baseline measurement as dependent variables, treatment, country, BG excursion, visit and treatment-by-visit interaction as fixed effects, baseline SMBG variable value as a covariate and participants as a random effect.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least 1 dose of study drug and had baseline and Week 26 body weight measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
kilogram (kg) | 2.31 [1.85 to 2.77] | 2.32 [1.84 to 2.79]

5. Secondary Outcome: Number of Hypoglycemic Events Baseline Through Week 26 (Incidence)
Description: A hypoglycemic event is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has a BG concentration of ≤ 70milligrams/deciliter [mg/dL (3.9 mmol/L)], even if it was not associated with signs, symptoms, or treatment consistent with current guidelines [American Diabetes Association (ADA) 2005].
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
events
  All Hypoglycemic Events | 568 | 583
  Severe Hypoglycemic Events | 0 | 1

6. Secondary Outcome: Insulin Dose at Week 26
Description: Insulin dose is the total daily dose including basal and prandial doses.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug and analyzed according to the assigned treatment regardless of study drug dose the participant received and had Week 26 insulin dose measurement.
Measure: Mean (Standard Deviation); unit: units of insulin per day (IU/day)
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
units of insulin per day (IU/day) | 40.02 (17.771) | 39.32 (17.991)

7. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG) at Week 26
Description: LS means were calculated by MMRM analysis using change from baseline in 1.5-AG variables at all post baseline measurement as dependent variables, treatment, country, BG excursion, visit and treatment-by-visit interaction as fixed effects, baseline SMBG variable value as a covariate and participants as a random effect.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least 1 dose of study drug and analyzed according to the assigned treatment regardless of study drug dose the participant received and had baseline and Week 26 1,5-AG measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: micrograms/milliliter (µg/mL)
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Number analyzed (Participants) | 207 | 196
micrograms/milliliter (µg/mL) | 4.24 [3.39 to 5.10] | 5.62 [4.74 to 6.51]

ADVERSE EVENTS:
Arm/Group | Insulin Lispro Mix25 | Insulin Lispro Mix50
Serious Adverse Events (participants affected / at risk) | 8/207 | 7/196
Other Adverse Events (participants affected / at risk) | 87/207 | 84/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Mix25 (N=207) | Insulin Lispro Mix50 (N=196)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro Mix25 (N=207) | Insulin Lispro Mix50 (N=196)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Arteriosclerotic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (6)
Dental caries (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Oesophageal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (2) | 0 (0)
Injection site induration (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (2)
Local swelling (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (4)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 28 (32) | 34 (42)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Endoscopy gastrointestinal (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 9 (9) | 12 (12)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 2 (2)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (16)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/131 (1) | 0/119 (0)
Menstruation delayed (Reproductive system and breast disorders) | 1/76 (1) | 0/77 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (2) | 2 (2)
Vocal cord nodule removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days